CLINICAL TRIAL: NCT00251329
Title: Phase II Neoadjuvant Trial of Docetaxel (Taxotere), Carboplatin, and Capecitabine (Xeloda) in the Treatment of Early Stage Locally Advanced and Inflammatory Breast Cancer
Brief Title: Docetaxel, Carboplatin, and Capecitabine as Treatment for Patients With Locally Advanced or Inflammatory Breast Cancer Before Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Research Network (Other)
Collaborators: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRN-004
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant; Breast Cancer; pCR; Capecitabine; Carboplatin; Docetaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

INTERVENTIONS:
Drug: neoadjuvant chemotherapy

SUMMARY:
The purpose of this study is to determine if this combination is safe and effective in this situation especially to increase the rate of pathological complete response (PCR). Women with large tumors and or lymph node involvement at the time of initial diagnosis may benefit from receiving chemotherapy prior to surgery to shrink the tumor and to decrease the amount of tumor involvement before surgery. If chemotherapy given before breast surgery is effective in decreasing the size of the tumor, breast conserving surgery (lumpectomy) may be possible. This new combination may be better tolerated than other commonly used regimens and, to date, appears to be at least as effective.

DETAILED DESCRIPTION:
Neoadjuvant (primary) chemotherapy is being used more frequently in locally advanced breast cancer in an effort to reduce the size of the primary tumor prior to surgery and to eliminate micrometastatic disease.Through previous studies, it has been shown that patients who receive neoadjuvant therapy demonstrate prolonged disease-free survival when compared to those who did not have a pCR at the time of surgery.

It is proven that docetaxel is the single most active drug in metastatic breast cancer treatment and therefore has sparked interest in its use in the neoadjuvant setting. There have been studies conducted using docetaxel either alone or in combination in this setting and in one particular study showed that patients treated with docetaxel after an anthracycline -containing regimen achieved at 34% pCR compared to only 16% with the anthracycline-containing regimen alone. This drugs low incidence of neutropenia when administered on a weekly schedule, plus its possible synergistic effects with carboplatin and capecitabine lead to its inclusion in this neoadjuvant protocol.

Carboplatin is an agent that has recently been integrated into the front line of breast cancer treatment due to its response rate and tolerability. This drug as well has warranted further investigation in the neoadjuvant setting and was combined with docetaxel in one trial for for locally advanced disease which showed a preliminary pCR of the breast and axilla of 30% and 80% respectively. Due to its tolerability, minimal toxicities, and impressive results as a single agent and in combination with docetaxel made carboplatin a reasonable drug of choice in this study.

The novel oral agent capecitabine is being used in this protocol because it has shown through study to significantly increase response rate, time to progression, and even overall survival when combined with docetaxel in the metastatic setting. As well, capecitabine behaves similarly to continuous 5-FU infusion which has shown success in several phase II neoadjuvant trials and essentially has led to its inclusion in this study. Capecitabine's anti-tumor activity, coupled with ease of administration, potential synergism with docetaxel and carboplatin, and non-overlapping toxicities justifies its inclusion in this investigational regimen.

ELIGIBILITY:
Inclusion Criteria:

* Women or men > 18 years old with histologically confirmed, by needle core biopsy (not FNA), locally advanced or inflammatory breast cancer.
* All patients must have either T2 lesion which is felt to be initially resectable only through mastectomy by the surgeon, or with a T3 N0-N2; T4 any N; or any T with N2 or N3 clinical evidence of disease. Stage 2 patients where breast conservation surgery is desired but impractical at diagnosis because of anticipated poor cosmetic outcome are eligible. Patients with inflammatory breast carcinoma and women with ipsilateral supraclavicular node involvement are eligible. Patients must have measurable disease defined as a breast lesion > 2 cm or with fixed or marked ipsilateral axillary nodes and/or ipsilateral internal mammary nodes.
* Pre-and Post-menopausal female and male patients are eligible. Women of childbearing potential must have a negative pregnancy test and, men and women must be willing to consent to using effective dual methods of contraception while on treatment and for three months thereafter.
* Life expectancy of greater than 6 months.
* Bone scan and CAT scan of chest and abdomen negative for metastatic disease

Exclusion Criteria:

* Patients with metastatic disease.
* Patients may not be receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection other than mild resolving cellulitis, symptomatic congestive heart failure (NYHA > Class 1), unstable angina pectoris, uncontrolled cardiac arrhythmia, known coronary artery disease, or psychiatric illness/social situations that would limit compliance with study requirements.
* Cancer other than breast primary within the last 5 years with the exception of surgically cured non-melanoma skin cancer or in situ carcinoma of the cervix.
* Women who are breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2003-05

PRIMARY OUTCOMES:
The primary objective of this study is to establish the pathological complete response rate (pCR) in the breast. The pCR is defined as the absence of invasive carcinoma.

SECONDARY OUTCOMES:
Establish pCR in breast and axillary lymph nodes
Establish pCR in axillary lymph nodes
Objective clinical response rate
Tolerability
Rate of breast conserving surgery
Time to disease progression
Local control rates

CONTACTS AND LOCATIONS:
Overall Officials: Sandra X Franco, MD, Principal Investigator — Cancer Research Network, Inc.
Locations (6):
- United States (6):
  - Baptist Cancer Institute, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Mount Sinai Comprehensice Cancer Center, Miami, Florida
  - Oncology /Hematology Associates of Florida, Miami, Florida
  - Cancer Research Network, Inc., Plantation, Florida
  - Sos/Acorn, Memphis, Tennessee